CLINICAL TRIAL: NCT02705404
Title: A Clinical Test for the Treatment of Multifocal Lung Cancers Using Genome
Brief Title: A Clinical Test for the Treatment of Multifocal Lung Cancers Using Genome Sequencing
Status: Terminated | Type: Observational
Why Stopped: Additional mechanisms/trials to enroll these patients exist and competed with the trial.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Marie Christine Aubry, MD, Principal Investigator, Mayo Clinic
Other Study IDs: 15-007961
Record Dates: First submitted 2016-02-22; First posted 2016-03-10 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Lung Neoplasms; Carcinoma Non-small-cell Lung
Keywords: multifocal; genetic; bronchoalveolar carcinoma; adenocarcinoma in situ; ground glass opacity; next generation sequencing
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma, Bronchiolo-Alveolar; Adenocarcinoma in Situ

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Biospecimen Retention: Samples With DNA — The patient will have some or all of the samples taken listed below:
  * Blood sample of 10 ml (2 teaspoons).
  * Up to two lung bronchoscopic or transbronchoscopic needle aspiration biopsies will be given to the research study during an already scheduled bronchoscopy. In addition at the time of the bronchoscopy a brushing or washing specimen could be collected for research.
  * A piece of lung or lymph node tissue taken at the time of the CT guided lung or lymph node biopsy will be given to the research study.
  * A piece of lung tumor tissue removed during surgery will be given to the research study.
  * If pleural fluid is removed as part of the procedure(s) and there is any fluid left after what is needed for your clinical care, it will be given to the research study.
  * DNA genome sequencing will be performed on the collected tissues, blood and fluid.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Multifocal Tissue Banking

SUMMARY:
The investigators are doing this research to see if they can use small tissue samples or fluid to develop a test that will determine if the tissue samples are related or not related to each other. The test will use the patient's DNA, which is part of their unique genetic material that carries the instructions for the body's development and function. Cancer can result from changes in a person's genetic material that causes cells to divide in an uncontrolled way and, sometimes, to travel to other organs. Currently, researchers and doctors know some of the genetic changes that can cause cancer, but they do not know all of the genetic changes that can cause cancer.

DETAILED DESCRIPTION:
A frequent clinical dilemma in lung cancer care is the management of multifocal lung cancers. The management decision is based on determining if multiple cancers represent true independent primary cancers or related metastasis. This determination is critical to the appropriate staging of the cancers and treatment. Indeed, this distinction represents the difference between aggressive local therapy with either surgery or radiation therapy for primary early stage lesions, or palliative chemotherapy or best supportive care with appropriate symptom management for advanced stage metastatic disease.

No existing pathologic or molecular test is currently capable of making the distinction between multiple independent lung primaries from metastatic disease with accuracy. The recent release of preliminary data from the NLST screening trial, suggesting survival benefit for screening high risk patients with CT scanning, will only increase the number of patients facing these treatment dilemmas. The research team has recently developed a test that allows this distinction with great accuracy. This test allows determination of lineage between two tumors using the identification of large genomic rearrangements using mate pair next generation sequencing (MP). The test has been developed using fresh frozen tissue from resected lung tumors and is currently being validated for a clinical test.

The investigators' goal is to develop the test using cytology and small biopsy specimens.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be > 18 years of age
* Presumed or known lung cancer.
* Undergoing bronchoscopy, CT guided lung biopsy, or lung resection as part of their clinical care at the Mayo Clinic Rochester.
* PFT's and other clinical determinates that show the subject is capable of tolerating a lung biopsy or resection.
* Non-pregnant and non-lactating. Women of child-bearing potential must have a negative urine or serum pregnancy test to participate in the study.
* Subject must be able to understand and willing to sign an IRB-approved informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic Rochester Patients
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Feasibility measured by being able to gather small samples from patients and having enough tissue to get results from the mate pair next generation sequencing. | 1 year
  Performance of the mate pair next generation sequencing lineage test on cytology and small biopsy specimens obtained as part of routine clinical practice, through either a bronchoscopic, CT-guided needle procedure, or lung resection as evidenced in receiving results from the sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Christine Aubry, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials